CLINICAL TRIAL: NCT03030729
Title: Macular Thickness Measurements Using RTOCT
Brief Title: Macular Thickness Measurements Using Retinal-thickness OCT
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: TLV-0025-16
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2017-01

CONDITIONS: Age-Related Macular Degeneration; Diabetic Retinopathy
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Intermediate AMD
- Advanced AMD
- DR without macular edema
- DR with macular edema

SUMMARY:
Comparison between retinal measurements, done by the RT (Retinal Thickness) imaging and a commercial OCT (Optical Coherence Tomography)

ELIGIBILITY:
Inclusion Criteria:

1. Ability and agreement to give informed consent (IC)
2. Diagnosis of AMD or DR in SE by OCT
3. Ability to undergo OCT scans

Exclusion Criteria:

1. AMD and DR in the same SE
2. Evidence of macular disease other than AMD or DME in SE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. AMD population - intermediate and advanced AMD (with active and non-active CNV)
  2. DR population. Patient with and without DME
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Comparison between retinal measurements, done by the RTOCT device and a commercial OCT | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sorasky Medical Center, Tel Aviv, Israel